CLINICAL TRIAL: NCT00793754
Title: Aspirin Statins Or Both For The Reduction Of Thrombin Generation In Diabetic People
Acronym: RATIONAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion GESICA (Other)
Responsible Party: Alejandro Macchia, Fundacion GESICA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Aspirin; Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention)
- 2 (Experimental): Aspirin 100 mg / day
  Interventions: Drug: Aspirin
- 3 (Experimental): Atorvastatin 40 mg / day
  Interventions: Drug: Atorvastatin
- 4 (Experimental): Aspirin 100 mg / day + Atorvastatin 40 mg / day
  Interventions: Drug: Aspirin + Atorvastatin

INTERVENTIONS:
Drug: Aspirin — 100 mg / day for 8 weeks
  Arms: 2
Drug: Atorvastatin — 40 mg / day for 8 weeks
  Arms: 3
Drug: Aspirin + Atorvastatin — Aspirin 100 mg / day + Atorvastatin 40 mg / day for 8 weeks
  Arms: 4

SUMMARY:
Despite formal recommendations, evidence of efficacy of aspirin in individuals with diabetes is scant and controversial. While the efficacy of aspirin versus placebo in patients with diabetes is currently under investigation in big randomized controlled trials, the putative additive effects of aspirin and statins in this population remain to be investigated. Moreover there are no data examining the pathophysiologic means by which aspirin with or without statins affects thrombosis in diabetic patients.

The aim of this trial is to evaluate the efficacy of low-dose aspirin (100 mg/daily), statins, both or neither for the reduction of thrombin generation. These preventive strategies will be evaluated on the top of the other strategies aimed at optimizing the care of diabetic patients in terms of metabolic control and control of the other cardiovascular risk factors.

DETAILED DESCRIPTION:
Despite the very high cardiovascular risk profile, evidence of efficacy of aspirin in individuals with diabetes is scant.

The meta-analysis on the efficacy of antiplatelet therapy involving a total of about 5,000 diabetic subjects indicates a non significant reduction in the risk of major cardiovascular events of 7%, compared with a reduction of 25% documented in secondary prevention studies.

Diabetes could represent a special case of aspirin resistance, although no specific studies have, to our knowledge, fully explored this hypothesis. The poor platelet responsiveness to aspirin has been recently proposed as a possible explanation of the failure of antiplatelet therapy to prevent cardiovascular events. The reduction in the aspirin activity in some patients is indicated by the failure in adequately suppressing thromboxane-A2 synthesis, as documented by the presence of high levels of its urinary metabolites.

The substantial lack of clear evidence is reflected by the low use of this drug in clinical practice; in fact, only 10% of diabetic patients are treated with aspirin for the prevention of cardiovascular events.

On the other hand, statins provide a similar efficacy for the prevention of major cardiovascular events in populations with and without diabetes.

It has been recently shown that platelet response to aspirin is linearly reduced with increasing cholesterol plasma levels. The presence of dyslipidemia, particularly common among diabetic patients, could thus be at least partially responsible for a lower efficacy of aspirin in this population. The concomitant use of statins could thus restore the normal platelet sensitivity to aspirin by reducing cholesterol levels

One additional reason to hypothesize a positive effect of statins in improving platelet response to aspirin is related to their anti-inflammatory properties

While the efficacy of aspirin versus placebo in patients with diabetes is currently under investigation, the additive effects of aspirin and statins in this population remain to be investigated. This aspect is of particular interest in the light of the existing debate regarding the need of multiple interventions to reduce total cardiovascular risk.

Given these premises, it is important to evaluate the effectiveness of aspirin use in primary prevention of cardiovascular events in association with statins therapy when included in a strategy of global risk control.

The RATIONAL Study will evaluate whether the combined use of aspirin (100 mg d) and statins (Atorvastatin 40 mg daily) is superior to the use of these single agents for the reduction of thrombin generation in patients with diabetes and without previous cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus treated with insulin or orl agents
* At least 50 years old

Exclusion Criteria:

* Previous cardiovascular events
* current or past (within last 30 days) treatment with aspirin
* current or past (within last 180 days) treatment with statins

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Thrombin generation | 8 weeks

SECONDARY OUTCOMES:
C-reactive protein | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Macchia, MD, Principal Investigator — Fundacion GESICA; Hernan Doval, MD, Principal Investigator — Fundacion GESICA; Juan J Fuselli, MD, Principal Investigator — Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno; Pablo D Comignani, MD, Principal Investigator — Hospital Aleman
Locations (1):
- Centro de Educación Médica e Investigaciones Clínicas (CEMIC), Buenos Aires, Argentina

REFERENCES:
- [Derived] Macchia A, Laffaye N, Comignani PD, Cornejo Pucci E, Igarzabal C, Scazziota AS, Herrera L, Mariani JA, Bragagnolo JC, Catalano H, Tognoni G, Nicolucci A. Statins but not aspirin reduce thrombotic risk assessed by thrombin generation in diabetic patients without cardiovascular events: the RATIONAL trial. PLoS One. 2012;7(3):e32894. doi: 10.1371/journal.pone.0032894. Epub 2012 Mar 28. PMID 22470429